CLINICAL TRIAL: NCT05066126
Title: Mixed Presentation of Content on Social Media and Its Relevant Impacts on Recall of Tobacco Related Information
Brief Title: Mixed Presentation on Social Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 849610
Record Dates: First submitted 2021-10-01; First posted 2021-10-04 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Tobacco Use; Tobacco Dependence
Keywords: Modified Risk Tobacco Products; Information Recall; Tobacco; Tobacco Use; Social Media
MeSH Terms: conditions — Tobacco Use; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two between-group conditions: either receiving a high mixed presentation of content in the social media feed (where the topic varies from post to post), or a low mix of presentation of content in the social media feed (where the topic does not vary).
  Additionally, two further between-subject groups will be created by independently examining effects among current and former smokers.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High-Mixed Presentation / Current Smoker (Experimental): Current smokers receive a social media feed with a high-mixed presentation of content.
  Interventions: Behavioral: Mixed-Presentation of Content
- Low-Mixed Presentation / Current Smoker (Experimental): Current smokers receive a social media feed with a low-mixed presentation of content.
  Interventions: Behavioral: Mixed-Presentation of Content
- High-Mixed Presentation / Former Smoker (Experimental): Former smokers receive a social media feed with a high-mixed presentation of content.
  Interventions: Behavioral: Mixed-Presentation of Content
- Low-Mixed Presentation / Former Smoker (Experimental): Former smokers receive a social media feed with a low-mixed presentation of content.
  Interventions: Behavioral: Mixed-Presentation of Content

INTERVENTIONS:
Behavioral: Mixed-Presentation of Content — Participants in the high-mixed presentation of content conditions will receive a social media feed that varies greatly between topics, so that each subsequent post is on a different topic. In the low-mixed presentation of content condition, participants will be shown posts on any given topic grouped together.

SUMMARY:
This study is to understand how the presentation of information on social media influences processing and recall of information, particularly in relation to modified risk tobacco products. Participants will see a social media site where either (a) the topic of discussion varies between each post or (b) posts on the same topic are grouped together. They will then be asked to recall information about the posts they saw on the site.

ELIGIBILITY:
Inclusion Criteria:

* Must be a current or former smoker

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Recall of precise information | During experiment
  Binary outcome as to whether the individual can recognize the specific text from a social media post as having appeared or not appeared on the social media site.
Recall of general information | During experiment
  Binary outcome as to whether the individual can recognize the content from a social media post as having appeared or not appeared on the social media site, but not necessarily the specific wording used.
Recall of source category | During experiment
  Binary outcome as to whether the individual can recognize the type of source (e.g. government/media) that presented a piece of information on the social media site.
Recall of precise source | During experiment
  Binary outcome as to whether the individual can recognize the exact source that presented a piece of information on the social media site.

SECONDARY OUTCOMES:
Attention paid during use of the site (self-report) | During experiment
  A series of questions pertaining attention paid during use of the social media site. These are then combined into a single self-report measure.
Attention paid during use of the site (behavioral) | During experiment
  Time spent consuming relevant posts on the social media site between conditions.
Attitude towards smoking cessation | During experiment
  Change in the interest in smoking between the pre- and post-test among current smokers. Measured with one self-report item.
Attitude towards novel tobacco products | During experiment
  Attitude/interest in trying alternative tobacco products (e.g. e-cigarettes, heated tobacco) in the post-test.
Belief of heated tobacco safety | During experiment
  Measure of how safe the individual believes heated tobacco is in comparison to cigarette use.

CONTACTS AND LOCATIONS:
Locations (1):
- Annenberg School for Communication, Philadelphia, Pennsylvania, United States